CLINICAL TRIAL: NCT04088461
Title: Effect of Linagliptin + Metformin on Glucose Metabolism and Pancreatic Beta Cell Function in Patients With Prediabetes Who do Not Achieve Normoglycemia After 12 Months of Treatment With Metformin Alone
Brief Title: Effect of Linagliptin + Metformin on Patients Who do Not Achieve Normoglucemia With Metformine
Acronym: RESCATHEME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Principal Investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEI-35-16
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Prediabetic State; Impaired Glucose Tolerance; Insulin Resistance
Keywords: Prediabetes; Insulin resistance; hyperglucemia
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Insulin Resistance | interventions — Linagliptin; Metformin; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin + Metformin and lifestyle (Experimental): Patients with impaired glucose tolerance randomly assigned to linagliptin 2.5 mg + metftormin 850 mg every 12 hours during 6 months.
  Interventions: Drug: Linagliptin / Metformin Oral Tablet
- Metformin (Active Comparator): Patients with impaired glucose tolerance randomly assigned to metftormin 850 mg every 12 hours during 6 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Linagliptin / Metformin Oral Tablet — Linagliptin 2.5 mg + Metformin 850 mg twice daily plus a lifestyle modifications program
  Other Names: Combined treatment
  Arms: Linagliptin + Metformin and lifestyle
Drug: Metformin — Metformin 850 mg twice daily plus lifestyle modifications program
  Other Names: Metformin alone
  Arms: Metformin

SUMMARY:
The goal of this protocol is to evaluate the effect of addhing linagliptin to patients with prediabetes who do not reverse to normoglycemia after 12 months of treatment with metformin alone. The duration of the study will be 6 months, and it is primarily a efficacy study. Main outcomes will be glucose levels during OGTT, insulin secretion and pancreatic beta cell function measured by the disposition index derived from the OGTT.

DETAILED DESCRIPTION:
Randomization and masking. Patients will be randomly assigned in a 1:1 ratio to receive linagliptin/metformin 2.5/850mg every 12 h + lifestyle modification program, or metformin 850mg every 12 h + lifestyle modification program during 6 months. Randomization will be performed using an electronic random numbers table by a Nutritionist not involved in the study. Participants and investigators involved in the patients follow-up and outcome measurements will be masked to treatment allocation during the entire study.

Patients will have a follow-up visit every month. Every appointment is about 30-45 minutes; medications tolerance and side effects will be recorded in every patients´ visit. Nutritional and physical activity assessment according to the patient´s weight will be performed by a Nutritionist every month. Monthly adherence to medications will be evaluated by pill counting; nutritional adherence and energy intake will be evaluated at 6 months by a food frequency questionnaire, and physical activity at 0 and 6 months. At basal and at 6 months patients will have an OGTT. Primary objective is to evaluate at 6 months glucose profile during OGTT, insulin secretion and pancreatic β-cell function by the OGTT DI, and regression to normoglycemia; T2D will be diagnosed and confirmed by at least two consecutive measurements of the same criteria: glycated haemoglobin ≥ 6.5 %, fasting glucose ≥ 126mg/dl, or 2 h glucose ≥ 200 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impaired glucose tolerance (2 h glucose between 140 - 199 mg / dL) that after 1 year of treatment with metformin at a dose of 1700 mg daily + lifestyle modifications don't achieve normoglycemia.
* Patients who accept to participate in the study and sign informed consent.

Exclusion Criteria:

* Patients with type 2 Diabetes diagnosted previuosly or detected during the OGTT
* Serum creatinine > 1.6 mg/dL
* Hypertriglyceridemia very high (>500 mg/dL)
* Pregnancy
* Systolic blood pressure > 180 mmHg or Diastolic blood pressure >105 mmHg (patients could be re-screened after blood pressure control)
* Excessive alcohol intake, acute or chronic
* Medications or medical conditions that affect glucose homeostasis (thiazides, beta blockers, glucocorticoids for systemic use, weight-reducing drugs or anorexigenics, Cushing's syndrom, Thyrotoxicosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Glucose levels during OGTT | 6 months
  Glucose levels during OGTT
Pancreatic beta cell function | 6 months
  Pancreatic beta cell function measured with the disposition index during OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado Mendoza, MDPhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez-Canales MFL, Salazar-Lopez SS, Farfan-Vazquez D, Martinez-Lopez YE, Gonzalez-Mena JN, Jimenez-Ceja LM, Vargas-Ortiz K, Evia-Viscarra ML, Montes de Oca-Loyola ML, Folli F, Aguilar-Garcia A, Guardado-Mendoza R. Effect of linagliptin on glucose metabolism and pancreatic beta cell function in patients with persistent prediabetes after metformin and lifestyle. Sci Rep. 2021 Apr 22;11(1):8750. doi: 10.1038/s41598-021-88108-8. PMID 33888772

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04088461/Prot_SAP_000.pdf